CLINICAL TRIAL: NCT06523322
Title: Culinary Medicine for Caregivers: Improving Pediatric Cancer Patient and Caregiver Outcomes Through Nutrition and Culinary Support
Brief Title: Culinary Medicine for Cancer Caregivers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Brandy-Joe Milliron, Associate Professor, Drexel University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-021869
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Pediatric Cancer; Caregiver Burden; Cancer, Treatment-Related; Nutrition Aspect of Cancer
Keywords: Culinary medicine; Nutrition; Cancer caregiver
MeSH Terms: conditions — Neoplasms; Caregiver Burden; Neoplasms, Second Primary

STUDY DESIGN:
Intervention Model Description: The 8-week Let's Cook Together program is intended to increase: caregiver knowledge of the benefits of a whole foods approach to eating; preparedness for caregiving; and caregiver self-efficacy for managing patients' nutrition-related side effects. The entire program will be delivered remotely. Caregivers will be recruited to participate in an 8-week remote culinary medicine intervention, including four remote synchronous culinary workshops (one 90-minute introductory event and three, 90-minute culinary/cooking sessions), and four bi-weekly caregiver coaching telephone calls (lasting 15-20 minutes).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Culinary Medicine plus Caregiver Coaching (Experimental): 8-week culinary medicine program, including 4 biweekly culinary medicine workshops and biweekly caregiver coaching.
  Interventions: Behavioral: Let's Cook Together

INTERVENTIONS:
Behavioral: Let's Cook Together — The 8-week Let's Cook Together program is intended to increase: caregiver knowledge of the benefits of a whole foods approach to eating; preparedness for caregiving; and caregiver self-efficacy for managing patients' nutrition-related side effects. The entire program will be delivered remotely. Caregivers will be recruited to participate in an 8-week remote culinary medicine intervention, including four remote synchronous culinary workshops (one 90-minute introductory event and three, 90-minute culinary/cooking sessions), and four bi-weekly caregiver coaching telephone calls (lasting 15-20 minutes).

SUMMARY:
Pediatric cancer and the therapies used in treatment can affect nutritional status, which can impact treatment tolerance, survival, and overall well-being. Poorly managed side effects can lead to long-term poor dietary habits. Caregivers who endure the psychosocial toll of these effects, also face risks to their own well-being. Prioritizing interventions that enhance caregivers' ability to provide quality care and improve long-term health is crucial. The primary aim of this study is to determine the feasibility and acceptability of an 8-week culinary medicine intervention with caregiver coaching for caregivers of children undergoing cancer treatment. The secondary aim is to estimate the effect of the intervention on caregiving preparedness, caregiver self-confidence for managing patient treatment side effects, eating-related distress, and dietary intake. In-depth interviews will explore participant experiences and perspectives on the feasibility and acceptability of the culinary nutrition program, and to inform interpretation of findings and future program refinement.

DETAILED DESCRIPTION:
Pediatric cancer and the therapies used in treatment can affect nutritional status, which can then impact treatment tolerance, survival, and overall well-being. Poorly managed side effects can lead to long-term poor dietary habits. Caregivers who endure the psychosocial toll of these effects, also face risks to their own well-being. Prioritizing interventions that enhance caregivers' ability to provide quality care and improve long-term health is crucial. Culinary medicine interventions have demonstrated efficacy in boosting cooking confidence and dietary quality as well as providing positive benefits to help with cancer treatment side effects. The investigators developed an 8-week culinary nutrition program incorporating caregiver coaching to enhance outcomes for pediatric cancer patients and their caregivers. Let's Cook Together aims to increase caregiver knowledge of a whole foods approach to eating, enhance preparedness for caregiving, and boost caregiver self-efficacy for managing side effects. Caregivers with children undergoing cancer treatment will be recruited from the Children's Hospital of Philadelphia. The program includes four remote cooking sessions led by a Medical Chef Educator and a Registered Dietitian Nutritionist, and bi-weekly coaching sessions to discuss caregiving goals, challenges, and problem-solving strategies. Written resources including nutrition education and recipes will be provided to all study participants. A single-arm mixed-methods feasibility study will assess the program's viability. Participants will undergo assessments at baseline, post-intervention, and three months post-intervention, with qualitative interviews post-intervention. The primary goal is to evaluate feasibility and acceptability, while secondary objectives include assessing preliminary efficacy on caregiving preparedness, caregiver self-efficacy, pediatric feeding behaviors, and dietary intake/behaviors. Results from the feasibility pilot, including qualitative feedback, will be used to guide the interpretation of findings, refine the study methodology and Let's Cook Together program, and inform the design of an adequately powered definitive trial. Findings may be of interest to a broad range of oncology and allied health professionals engaged in supportive care for families experiencing cancer treatment.

ELIGIBILITY:
*Please note the above age limit and 'accepts health volunteers' specifications are related to the caregiver as the participant. Additional age limit criteria for patient is listed below. All caregivers will be providing care for a child undergoing current cancer treatment.

Inclusion Criteria, Patient:

* Receiving active cancer treatment for a liquid or solid cancer diagnosis
* At least 4-17 years of age
* English-speaking
* Taking >50% intake orally
* Approved to participate by both their oncologist and registered dietitian nutritionist

Exclusion Criteria, Patient:

* Undergoing bone marrow transplantation
* Receiving active cancer treatment for a brain tumor

Inclusion Criteria, Caregiver:

* Caregiver (parent or legal guardian) of a child who meets the inclusion and exclusion criteria for patients, above
* Can read and speak English
* Has access to a computer (i.e., tablet, laptop, desktop computer) and internet
* Is at least 18 years of age
* Has the ability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-25 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention as assessed by participant session attendance, assessment completion, and participant retention. | During the intervention; immediately after the intervention; and 3-months after the intervention
  Objective metrics will be used to determine feasibility, including the number of participants enrolled per month of recruitment, the percent of participants who provide assessment data at 8 weeks, and the proportion of retained participants who provide valid data for each assessment task. The percent of participants who attend all sessions and complete all assessments will be used as a metric for feasibility.
Acceptability of the intervention as assessed by comprehension of intervention content, personal relevance, and appropriate information volume. | During the intervention; immediately after the intervention; and 3-months after the intervention
  Acceptability will be measured along a 5-point Likert scale to questions that ask whether the culinary medicine information was easy to understand, personally relevant, and whether the amount of information presented was appropriate. Intervention acceptability will be expressed as the percent of participants who rate each of the previous domains as 'agree' or 'strongly agree.'
Usage of the intervention as assessed by the number of recipes used. | During the intervention; immediately after the intervention; and 3-months after the intervention
  Usage will be measured according to the number of recipes used.
Usability of the intervention as assessed by ease of use and plan for continued use. | During the intervention; immediately after the intervention; and 3-months after the intervention
  Usability will be measured along a 5-point Likert scale to questions that ask participants the extent to which the recipes were easy to use and plan for continued use. Intervention usability will be expressed as the percent of participants who rate each of the previous domains as 'agree' or 'strongly agree.'
Perceived usefulness as assessed by the extent to which the session was useful in helping participants to increase their confidence, overcome barriers, and increase the support they receive. | During the intervention; immediately after the intervention; and 3-months after the intervention
  Perceived usefulness will be measured along a 5-point Likert scale to questions ask the extent to which the session was useful in helping participants to increase their confidence, overcome barriers, and increase the support they receive. Perceived usefulness will be expressed as the percent of participants who rate each of the previous domains as 'agree' or 'strongly agree.'

SECONDARY OUTCOMES:
Change from baseline in preparedness for caregiving as assessed by the Preparedness for Caregiving Scale. | Baseline; immediately after the intervention; and 3-months after the intervention
  Caregiving Preparedness will be assessed using the Preparedness for Caregiving Scale, an 8-item survey that assesses caregivers' readiness to provide care for the patient and includes multiple domains of caregiving, such as providing physical care and emotional support. Answers are given using a five-point Likert-type scale (answers range from 'not at all prepared' [0] to 'very well prepared' [4]). Overall preparedness will be determined by calculating the average of the eight survey items. Higher scores indicate better preparedness.
Change from baseline in caregiver self-efficacy to manage treatment-related side effects a assessed by the Caregiver Self-Efficacy for Management of Treatment Side Effects survey | Baseline; immediately after the intervention; and 3-months after the intervention
  Caregiver self-efficacy will be assessed using the Caregiver Self-Efficacy for Management of Treatment Side Effects survey, a 16-item survey to assess caregiver confidence in their abilities to manage cancer treatment side effects. Item ratings range from 10 (very uncertain) to 100 (very certain), where higher scores indicate greater self-efficacy. Overall self-efficacy is calculated using the mean of the 16 items. Additional scores will be calculated for self-efficacy for managing function-related side effects, pain, and 'other' side effects. 'Other' side effects include fatigue, lack of appetite, nausea, shortness of breath, feeling blue and frustration.
Change from baseline in caregiver eating-related distress as assessed by the Behavioral Pediatrics Feeding Assessment Scale. | Baseline; immediately after the intervention; and 3-months after the intervention
  The Behavioral Pediatrics Feeding Assessment Scale (BPFAS) is a 35-item scale assesses behaviors associated with poor nutritional intake. The first 25 questions focus on the child's behavior and the next 10 questions focus on parental feelings or strategies for dealing with eating problems. Each item displays a descriptive phrase for which the caregiver is asked to rate how often the behavior occurs on a 5-point Likert scale from "never" to "always" and whether or not the caregiver considered the behavior to be a problem (yes" or "no"). Higher scores indicate greater eating-related distress.
Change from baseline in caregiver dietary intake as assessed by the Inflammatory Diet Index. | Baseline; immediately after the intervention; and 3-months after the intervention
  Dietary intake will be collected and analyzed using the Diet History Questionnaire III (DHQ III), developed by the National Cancer Institute, Bethesda, MD. The DHQ III is a freely available, web-based food frequency questionnaire for use with adults 19 or more years of age. The DHQ III consists of 135 food and beverage items and 26 dietary supplement questions and can be used to examine dietary intake over the previous month. Participant responses to the DHW III will be scored for the inflammatory index of their diet using the Dietary Inflammatory Index (DII). Scores range from -8.87 to 7.98. Higher scores indicate greater inflammatory property of diet.
Change from baseline in patient dietary intake (food groups, macronutrient, micronutrient, and caloric intake) as assessed by the Automated Self-Administered 24-hour Dietary Assessment Tool | Baseline; immediately after the intervention; and 3-months after the intervention
  Caregivers will complete the Automated Self-Administered 24-hour Dietary Assessment Tool (ASA24) on behalf of the patient (their child) to collect information on dietary patterns and total caloric intake. ASA24 is an electronic-based dietary recall that is available free of charge through the National Cancer Institute.

OTHER OUTCOMES:
Participant experiences and perspectives on the culinary medicine program as assessed through qualitative data (in-depth interviews) | Immediately after the intervention; 3-months after the intervention
  In-depth interviews with caregivers will be conducted to explore their experiences and perspectives on the culinary medicine program to inform interpretation of findings and scale-up. For example, interviews will explore factors that hinder or facilitate use of recipes provided and strategies described during classes and will explore participants' interest in continued use of recipes and strategies as a preliminary indicator of program engagement and dissemination potential.

REFERENCES:
- [Derived] Milliron BJ, Mountain P, Salman K, Longo G, Schlechter H, Deutsch JM, Jubelirer T. Culinary medicine for caregivers: protocol for a mixed-methods feasibility study to improve pediatric cancer patient and caregiver outcomes through nutrition and culinary support. Pilot Feasibility Stud. 2025 Sep 30;11(1):120. doi: 10.1186/s40814-025-01703-8. PMID 41029472